CLINICAL TRIAL: NCT04839835
Title: The Effect of Art Design in the Chemotherapy Waiting Room on the Anxiety of Patients Who Will Receive Chemotherapy for the First Time
Brief Title: Anxiety on the First Day of Chemotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Asoc. Prof. Erdoğan Selçuk Şeber, Asoc. Prof., Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: waitingroom
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Anxiety
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard waiting room (No Intervention): standard chemoterapy waiting room
- waiting room enriched with art objects (Experimental): waiting room enriched with music, paintings and artificial plants
  Interventions: Other: waiting room enriched with music, paintings and artificial plants

INTERVENTIONS:
Other: waiting room enriched with music, paintings and artificial plants — waiting room enriched with music, paintings and artificial plants
  Arms: waiting room enriched with art objects

SUMMARY:
investigating chemotherapy anxieties

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women in the world, and it is the first in cancer-related deaths in women all over the world. In the treatment of breast cancer, in addition to surgery, patients with advanced stage or high risk of recurrence receive neoadjuvant and adjuvant chemotherapy treatments. This period starts with 3 months and extends according to the treatment protocols it will receive.

Since the first diagnosis of breast cancer, it has psychological effects such as intense stress, decrease in quality of life and anxiety as well as physical effects on patients. The time spent in the "waiting room" while patients are examined and receiving treatment before chemotherapy inevitably has an effect on their anxiety.

In this study; It was aimed to investigate the effects of environmental factors in waiting rooms on patients' anxiety.

ELIGIBILITY:
Inclusion Criteria:

* to receive chemotherapy for breast cancer for the first time
* give consent for the study

Exclusion Criteria:

* not approving to participate in the study

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-03-03 (Estimated)

PRIMARY OUTCOMES:
anxiety and stress measurements | 60-120 minutes
  The State-Trait Anxiety Inventory (STAI) - Measuring anxiety with the Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Locations (1):
- Tekirdağ Namık Kemal ÜNiversitesi, Tekirdağ, Turkey (Türkiye)